CLINICAL TRIAL: NCT02704468
Title: FGF21 Can Help Predicting Arterial Stiffness Measured by Cardio-ankle Vascular Index in Renal Transplant Patients
Acronym: CAVIFGF21
Status: Completed | Type: Observational
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associated Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Other Study IDs: 085/58
Record Dates: First submitted 2016-02-29; First posted 2016-03-10 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Vascular Stiffness
Keywords: CAVI; FGF-21; arterial stiffness; renal transplant
MeSH Terms: interventions — fibroblast growth factor 21

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CAVI and FGF-21: renal transplant patients for more than 1 month measured FGF-21 and CAVI
  Interventions: Other: CAVI and FGF-21

INTERVENTIONS:
Other: CAVI and FGF-21 — FGf-21 and CAVI was measured in renal transplant patients group and study correlation with arterial stiffness

SUMMARY:
Chronic kidney disease(CKD) patients have high incidence of coronary artery problems event after renal transplantation. And remain a major cause of mortality. The major risk marker is arterial stiffness. The cardio-ankle vascular index (CAVI) is a new index of overall stiffness and can estimated the risk of atherosclerosis.

Fibroblast growth factor 21 (FGF-21) is a metabolic regulator that plays important role in cardiac remodeling elevated FGF-21 have been reported in coronary heart disease or carotid artery plaque and could be biomarkers for atherosclerosis disease Investigators aimed to study the association between CAVI and FGF-21 and their relations to various parameters that can contribute to cardiovascular disease eg. homocysteine Echocardiogram findings and other traditional basic factors.

DETAILED DESCRIPTION:
A total of 90 participants who underwent renal transplant were included in the study. The following measures were done and laboratory data were collected. CAVI, Ecchocariogram, Homocysteine, Hs-CRP, Carotid IMT, FGF-21, Medication after renal transplantation, incidence of cardiovascular disease correlation between categorical data was done by using Pearson's correlation test and multiple regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant patients patients for more than 1 month

Exclusion Criteria:

* who had contraindication for CAVI
* current smoker
* eGFR <15 ml/min/173
* cardiac arrthymia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: renal transplant pateints for more than 1 month
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
association between CAVI and FGF-21 with arterial stiffness in renal transplant patients | 1 month
  cross sectional study

SECONDARY OUTCOMES:
association between Hs-CRP,Homocystein with CAVI | 1 month
  cross sectional study

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, M.D., Study Director — Bangkok metropolitan administration medical college of vajira hospital
Locations (1):
- Bangkok metropolitan administraiton of vajira hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data about CAVI and FGF 21

REFERENCES:
- [Background] Sarnak MJ, Levey AS, Schoolwerth AC, Coresh J, Culleton B, Hamm LL, McCullough PA, Kasiske BL, Kelepouris E, Klag MJ, Parfrey P, Pfeffer M, Raij L, Spinosa DJ, Wilson PW; American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Kidney disease as a risk factor for development of cardiovascular disease: a statement from the American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Circulation. 2003 Oct 28;108(17):2154-69. doi: 10.1161/01.CIR.0000095676.90936.80. No abstract available. PMID 14581387
- [Background] An SY, Lee MS, Yi SA, Ha ES, Han SJ, Kim HJ, Kim DJ, Lee KW. Serum fibroblast growth factor 21 was elevated in subjects with type 2 diabetes mellitus and was associated with the presence of carotid artery plaques. Diabetes Res Clin Pract. 2012 May;96(2):196-203. doi: 10.1016/j.diabres.2012.01.004. Epub 2012 Jan 30. PMID 22293928
- [Background] Verbeke F, Marechal C, Van Laecke S, Van Biesen W, Devuyst O, Van Bortel LM, Jadoul M, Vanholder R. Aortic stiffness and central wave reflections predict outcome in renal transplant recipients. Hypertension. 2011 Nov;58(5):833-8. doi: 10.1161/HYPERTENSIONAHA.111.176594. Epub 2011 Sep 6. PMID 21896935
- [Background] Khoshdel AR, Carney SL. Arterial stiffness in kidney transplant recipients: an overview of methodology and applications. Urol J. 2008 Winter;5(1):3-14. PMID 18454420
- [Background] Stehouwer CD, Henry RM, Ferreira I. Arterial stiffness in diabetes and the metabolic syndrome: a pathway to cardiovascular disease. Diabetologia. 2008 Apr;51(4):527-39. doi: 10.1007/s00125-007-0918-3. Epub 2008 Feb 1. PMID 18239908
- [Background] Sun CK. Cardio-ankle vascular index (CAVI) as an indicator of arterial stiffness. Integr Blood Press Control. 2013 Apr 30;6:27-38. doi: 10.2147/IBPC.S34423. Print 2013. PMID 23667317
- [Background] Kim KJ, Lee BW, Kim HM, Shin JY, Kang ES, Cha BS, Lee EJ, Lim SK, Lee HC. Associations between cardio-ankle vascular index and microvascular complications in type 2 diabetes mellitus patients. J Atheroscler Thromb. 2011;18(4):328-36. doi: 10.5551/jat.5983. Epub 2011 Jan 6. PMID 21224525
- [Background] Takaki A, Ogawa H, Wakeyama T, Iwami T, Kimura M, Hadano Y, Matsuda S, Miyazaki Y, Matsuda T, Hiratsuka A, Matsuzaki M. Cardio-ankle vascular index is a new noninvasive parameter of arterial stiffness. Circ J. 2007 Nov;71(11):1710-4. doi: 10.1253/circj.71.1710. PMID 17965489
- [Background] Hayashi K, Sato M, Niimi H, Handa H, Moritake K. [Analysis of the constitutive laws of the vascular wall by finite deformation theory]. Iyodenshi To Seitai Kogaku. 1975 Oct;13(5):293-8. No abstract available. Japanese. PMID 1240535
- [Background] KOTANI, K.; REMALEY, A. T. Cardio-AnkleVascular Index (CAVI) and its Potential Clinical Implications for Cardiovascular Disease. CardiolPharmacol, 2013, 2: 108.
- [Background] Otsuka K, Fukuda S, Shimada K, Suzuki K, Nakanishi K, Yoshiyama M, Yoshikawa J. Serial assessment of arterial stiffness by cardio-ankle vascular index for prediction of future cardiovascular events in patients with coronary artery disease. Hypertens Res. 2014 Nov;37(11):1014-20. doi: 10.1038/hr.2014.116. Epub 2014 Jul 10. PMID 25007768
- [Background] Dobsak P, Soska V, Sochor O, Jarkovsky J, Novakova M, Homolka M, Soucek M, Palanova P, Lopez-Jimenez F, Shirai K. Increased cardio-ankle vascular index in hyperlipidemic patients without diabetes or hypertension. J Atheroscler Thromb. 2015;22(3):272-83. doi: 10.5551/jat.24851. Epub 2014 Oct 22. PMID 25342382
- [Background] Shirai K, Hiruta N, Song M, Kurosu T, Suzuki J, Tomaru T, Miyashita Y, Saiki A, Takahashi M, Suzuki K, Takata M. Cardio-ankle vascular index (CAVI) as a novel indicator of arterial stiffness: theory, evidence and perspectives. J Atheroscler Thromb. 2011;18(11):924-38. doi: 10.5551/jat.7716. Epub 2011 May 31. PMID 21628839
- [Background] Cheng HM, Chuang SY, Sung SH, Yu WC, Pearson A, Lakatta EG, Pan WH, Chen CH. Derivation and validation of diagnostic thresholds for central blood pressure measurements based on long-term cardiovascular risks. J Am Coll Cardiol. 2013 Nov 5;62(19):1780-7. doi: 10.1016/j.jacc.2013.06.029. Epub 2013 Jul 10. PMID 23850921
- [Background] Jin K, LaFevre-Bernt M, Sun Y, Chen S, Gafni J, Crippen D, Logvinova A, Ross CA, Greenberg DA, Ellerby LM. FGF-2 promotes neurogenesis and neuroprotection and prolongs survival in a transgenic mouse model of Huntington's disease. Proc Natl Acad Sci U S A. 2005 Dec 13;102(50):18189-94. doi: 10.1073/pnas.0506375102. Epub 2005 Dec 2. PMID 16326808
- [Background] Kharitonenkov A, Shiyanova TL, Koester A, Ford AM, Micanovic R, Galbreath EJ, Sandusky GE, Hammond LJ, Moyers JS, Owens RA, Gromada J, Brozinick JT, Hawkins ED, Wroblewski VJ, Li DS, Mehrbod F, Jaskunas SR, Shanafelt AB. FGF-21 as a novel metabolic regulator. J Clin Invest. 2005 Jun;115(6):1627-35. doi: 10.1172/JCI23606. Epub 2005 May 2. PMID 15902306
- [Background] Coskun T, Bina HA, Schneider MA, Dunbar JD, Hu CC, Chen Y, Moller DE, Kharitonenkov A. Fibroblast growth factor 21 corrects obesity in mice. Endocrinology. 2008 Dec;149(12):6018-27. doi: 10.1210/en.2008-0816. Epub 2008 Aug 7. PMID 18687777
- [Background] Kharitonenkov A, Wroblewski VJ, Koester A, Chen YF, Clutinger CK, Tigno XT, Hansen BC, Shanafelt AB, Etgen GJ. The metabolic state of diabetic monkeys is regulated by fibroblast growth factor-21. Endocrinology. 2007 Feb;148(2):774-81. doi: 10.1210/en.2006-1168. Epub 2006 Oct 26. PMID 17068132
- [Background] Ong KL, Januszewski AS, O'Connell R, Jenkins AJ, Xu A, Sullivan DR, Barter PJ, Hung WT, Scott RS, Taskinen MR, Keech AC, Rye KA. The relationship of fibroblast growth factor 21 with cardiovascular outcome events in the Fenofibrate Intervention and Event Lowering in Diabetes study. Diabetologia. 2015 Mar;58(3):464-73. doi: 10.1007/s00125-014-3458-7. Epub 2014 Nov 26. PMID 25425220
- [Background] Lin Z, Wu Z, Yin X, Liu Y, Yan X, Lin S, Xiao J, Wang X, Feng W, Li X. Serum levels of FGF-21 are increased in coronary heart disease patients and are independently associated with adverse lipid profile. PLoS One. 2010 Dec 29;5(12):e15534. doi: 10.1371/journal.pone.0015534. PMID 21206918
- [Background] Mirza MA, Hansen T, Johansson L, Ahlstrom H, Larsson A, Lind L, Larsson TE. Relationship between circulating FGF23 and total body atherosclerosis in the community. Nephrol Dial Transplant. 2009 Oct;24(10):3125-31. doi: 10.1093/ndt/gfp205. Epub 2009 May 9. PMID 19429932
- [Background] Lee Y, Lim S, Hong ES, Kim JH, Moon MK, Chun EJ, Choi SI, Kim YB, Park YJ, Park KS, Jang HC, Choi SH. Serum FGF21 concentration is associated with hypertriglyceridaemia, hyperinsulinaemia and pericardial fat accumulation, independently of obesity, but not with current coronary artery status. Clin Endocrinol (Oxf). 2014 Jan;80(1):57-64. doi: 10.1111/cen.12134. Epub 2013 May 6. PMID 23278761
- [Background] Mahabadi AA, Massaro JM, Rosito GA, Levy D, Murabito JM, Wolf PA, O'Donnell CJ, Fox CS, Hoffmann U. Association of pericardial fat, intrathoracic fat, and visceral abdominal fat with cardiovascular disease burden: the Framingham Heart Study. Eur Heart J. 2009 Apr;30(7):850-6. doi: 10.1093/eurheartj/ehn573. Epub 2009 Jan 9. PMID 19136488
- [Background] Chow WS, Xu A, Woo YC, Tso AW, Cheung SC, Fong CH, Tse HF, Chau MT, Cheung BM, Lam KS. Serum fibroblast growth factor-21 levels are associated with carotid atherosclerosis independent of established cardiovascular risk factors. Arterioscler Thromb Vasc Biol. 2013 Oct;33(10):2454-9. doi: 10.1161/ATVBAHA.113.301599. Epub 2013 Jul 25. PMID 23887638
- [Background] Semba RD, Crasto C, Strait J, Sun K, Schaumberg DA, Ferrucci L. Elevated serum fibroblast growth factor 21 is associated with hypertension in community-dwelling adults. J Hum Hypertens. 2013 Jun;27(6):397-9. doi: 10.1038/jhh.2012.52. Epub 2012 Nov 29. PMID 23190795
- [Background] Chen YC, Lee MC, Lee CJ, Ho GJ, Yin WY, Chang YJ, Hsu BG. N-terminal pro-B-type natriuretic peptide is associated with arterial stiffness measured using the cardio-ankle vascular index in renal transplant recipients. J Atheroscler Thromb. 2013;20(7):646-53. doi: 10.5551/jat.17780. Epub 2013 May 10. PMID 23665842
- [Background] Deo R, Shou H, Soliman EZ, Yang W, Arkin JM, Zhang X, Townsend RR, Go AS, Shlipak MG, Feldman HI. Electrocardiographic Measures and Prediction of Cardiovascular and Noncardiovascular Death in CKD. J Am Soc Nephrol. 2016 Feb;27(2):559-69. doi: 10.1681/ASN.2014101045. Epub 2015 Jul 9. PMID 26160896